CLINICAL TRIAL: NCT06321549
Title: Shifting Strategic Approach in Breast Reconstruction Using Free DIEP Flap Along With The Paradigm Shifting of Mastectomy Technique
Brief Title: New Era of DIEP With Minimally Invasive Mastectomy
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Ju Huang, Associate Professor, Chang Gung Memorial Hospital
Other Study IDs: 202201562B0
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Breast Reconstruction; Mastectomy; Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Individuals who underwent surgery prior to November 2018
- Group B: Individuals who underwent surgery after November 2018
  Interventions: Other: The reference point of minimally invasive mastectomy procedure conducted

INTERVENTIONS:
Other: The reference point of minimally invasive mastectomy procedure conducted — November 2018 as a temporal reference point was predicated on the milestone of the medical center's inaugural minimally invasive mastectomy procedure conducted
  Groups: Group B

SUMMARY:
The free deep inferior epigastric artery perforator (DIEP) flap is the gold standard in autologous breast reconstruction. Asian patients often present with a smaller body mass index with relatively insufficient tissue. To restore appropriate symmetry, a larger flap inset ratio must be transferred. Supercharging of the second vein or inclusion of bilateral pedicle is commonly required. Current paradigm shifts in mastectomy has also resulted in more minimally invasive surgeries (MIS) espousing smaller lateral incisions, leading to a significant change in available recipient vessels. This study aimed to demonstrate our experience in changing strategies of DIEP flaps following the evolution of mastectomy techniques.

Between October 2008 and March 2022, retrospective data was gathered for 278 patients who underwent breast reconstruction surgery utilizing DIEP flaps by a single plastic surgeon. These patients were divided into two distinct groups based on their operation dates, with November 2018 marking a pivotal moment when the first MIS was introduced.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent breast reconstruction procedures with DIEP flaps from October 2008 to March 2022.
* Patients who have a minimum follow-up duration of six months post-reconstruction.

Exclusion Criteria:

* Patients who did not meet the six-month follow-up duration was excluded from the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent breast reconstruction procedures with DIEP flaps from October 2008 to March 2022 from a single experienced reconstructive surgeon's practice at a medical institution.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Endoscopy mastectomy | Post-operative day 0
Robotic mastectomy | Post-operative day 0
Incision | Post-operative day 0
Usage of SIEV | Post-operative day 0
Inclusion of bipedicle | Post-operative day 0
Location of recipient artery/vein | Post-operative day 0
Recipient artery/vein selection | Post-operative day 0

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Ju Huang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin TE, Wong AW, Cheong DC, Kuo WL, Tsai HP, Huang JJ. Strategically shifting paradigms: the new era of DIEP flaps with minimally invasive mastectomy: a retrospective cross-sectional study. BMC Cancer. 2024 Aug 30;24(1):1072. doi: 10.1186/s12885-024-12846-x. PMID 39210299